CLINICAL TRIAL: NCT02829905
Title: Women's Experiences of Mammography: Quantitative Evaluation
Acronym: WEM-Quant
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); University of St Andrews (Other)
Responsible Party: Principal Investigator, Patsy Whelehan, Senior Research Radiographer, University of Dundee
Other Study IDs: 2016ON15
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: mass screening; patient satisfaction; radiography; mammography
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study will develop, validate and pilot measures to assess quality of experiences of mammography. Pilot data collection and analysis will investigate modifiable factors most important in determining quality of patient experiences of mammography.

DETAILED DESCRIPTION:
While instruments to measure experiences of breast screening and mammography have been developed in the past, there is none which (a) concentrates in depth on the experience of the examination itself, (b) includes detailed breast positioning variables, (c) has been designed based on robust and transparent qualitative evidence, and (d) has been validated in a UK breast setting. Such a tool is needed to inform the design, development and testing of interventions to improve experiences of mammography. This is an important goal because many women are deterred from future breast screening by poor mammography experiences. Furthermore, regular client satisfaction surveys are required by the UK national breast screening programmes but there is no standard, validated measure in place.

The aim of this project is to develop, and obtain evidence for the validity of, a comprehensive toolkit of measures to evaluate experiences of mammography. The measures will be capable of assessing the quality of experiences of mammography and identifying modifiable predictors thereof. The investigators will pilot the measures in a sample of women attending for NHS breast screening. The resulting data will be used as the basis for building a statistical analysis model, for further validation of the measures, and for producing preliminary findings on what they are intended to measure.

Items generated from the investigators recent qualitative study will be combined with items from existing literature and with novel image-based metrics to draft comprehensive measures of women's mammography experiences. Questionnaires will capture 1. relevant modifiable potential determinants of overall quality of experience, such as the mammographer's ability to put the client at ease, 2. key potential confounding variables (e.g. client physical characteristics such as mobility problems or breast tenderness), and 3. outcome variables representing or postulated to contribute to overall quality of experience, including pain from the mammogram. Questionnaire development will follow established methods, including testing for face and content validity with a sample of field experts and of the target population, and checking for question design errors - such as leading questions - by a member of the team experienced in questionnaire construction. The draft questionnaires will be cognitively tested for understandability and acceptability with a small sample of women eligible for breast screening, and refined before administration to a larger sample of women attending for screening mammography. The questionnaire data will be incorporated into a statistical analysis model along with additional data which the investigators will extract from participants' mammographic images as follows.

The mammographic images will be examined for variables which may affect the client experience. These will include e.g. the compression force applied to the breast tissue during mammography, and features of the breast positioning technique. Thus, the measurement toolkit will have multiple parts. The investigators expect it to be capable of rigorous routine service and performance evaluation in mammography, of identifying what nature of interventions are needed to improve mammography experiences, and of evaluating the effectiveness of such interventions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for NHS breast screening
* Able to speak and write English.

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women eligible for population-based breast screening in the UK, i.e. aged 47+
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with mammography experience | Immediate
  11-point NRS

SECONDARY OUTCOMES:
Pain from mammography | Immediate
  11-point NRS
Intention to re-attend for mammography screening | Immediate
  11-point NRS

CONTACTS AND LOCATIONS:
Overall Officials: Patsy Whelehan, MSc, Principal Investigator — University of Dundee and NHS Tayside
Locations (1):
- Ninewells Hospital, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Applications considered on case by case basis.